CLINICAL TRIAL: NCT03504722
Title: Evaluating the Feasibility of Recovery Through Engagement With Shelter Canines, Understanding, and Exposure (RESCUE): An Adjunctive Human Animal Interaction (HAI)-Based Intervention for Veterans With PTSD
Brief Title: Evaluating the Feasibility of RESCUE: An Adjunctive HAI-Based Intervention for Veterans With PTSD
Acronym: RESCUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charleston Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH-15-1-0087
Record Dates: First submitted 2017-05-02; First posted 2018-04-20 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESCUE+PE (Experimental): RESCUE is designed to adapt to individualized needs based on each veteran's performance. The volunteer training consists of weekly sessions lasting 90 minutes each and occurring at area Society for the Prevention of Cruelty to Animals (SPCA) facilities.All veterans will receive individualized, evidence-based prolonged exposure therapy. Foa's PE protocol will be used given consensus statements indicating that exposure therapy is currently the most appropriate psychotherapy for PTSD.
  Interventions: Behavioral: RESCUE; Behavioral: Prolonged Exposure
- PE+delayed RESCUE (Active Comparator): All veterans will receive individualized, evidence-based prolonged exposure therapy. Foa's PE protocol will be used given consensus statements indicating that exposure therapy is currently the most appropriate psychotherapy for PTSD.
  Interventions: Behavioral: Prolonged Exposure

INTERVENTIONS:
Behavioral: RESCUE — RESCUE is designed to adapt to individualized needs based on each veteran's performance. The volunteer training consists of weekly sessions lasting 90 minutes each and occurring at area SPCA facilities. The logistics of the training sessions will be facilitated by study staff, with SPCA animal behaviorists and professionals conducting the training program identical to the program that they use for their general volunteer training. During volunteer sessions, the veteran learns behavioral techniques for training non-aggressive dogs through didactic instruction followed by demonstration and supervised practice. The animal socialization component of the RESCUE volunteer sessions are comprised of the SPCAs current training program, which is designed developmentally such that early training focuses on general topics (safety, basic handling skills) and later training builds on previously learned skills through successive approximation within each individual's zone of proximal development.
  Arms: RESCUE+PE
Behavioral: Prolonged Exposure — All veterans will receive individualized, evidence-based prolonged exposure therapy. Foa's PE protocol will be used given consensus statements indicating that exposure therapy is currently the most appropriate psychotherapy for PTSD. Study therapists are already trained clinicians through the VA's PE certification process and will receive weekly supervision for all cases from the PI, who is a national Prolonged Exposure trainer.
  Other Names: PE

SUMMARY:
To develop and pilot test feasibility, acceptability, and efficacy of an adjunct intervention for use with Empirically Based Treatments (EBT) for posttraumatic stress disorder (PTSD) in order to increase treatment engagement, treatment completion, and improve treatment response regarding emotional numbing symptoms. Recovery through Engagement with Shelter Canines, Understanding, and Exposure (RESCUE), is an adjunctive, Human Animal Interaction (HAI) intervention that will be developed for integration into Prolonged Exposure (PE) treatment. Feasibility, acceptability, and initial efficacy testing of the experimental treatment condition will be conducted in a pilot crossover randomized controlled trial (RCT) conducted with 75 veterans with PTSD randomly assigned to RESCUE delivered with PE (RESCUE+PE) or to standard PE initiation (PE + delayed RESCUE).

ELIGIBILITY:
Inclusion Criteria:

1. Veterans with a principal Diagnostic and Statistical Manual-5th edition (DSM-5) PTSD diagnosis (via CAPS) stemming from a Criterion A event.
2. Men or women aged 18 to 64 inclusive.
3. Given that individuals with PTSD often have comorbid psychiatric disorders, participants with comorbid depressive, anxiety, substance use disorders, and personality disorders other than Antisocial Personality Disorder will be included as long as PTSD is the primary disorder
4. Individuals with the ability to comprehend and satisfactorily comply with protocol requirements and who sign the written informed consent given prior to entering any study procedure

Exclusion Criteria:

1. Individuals with active substance use disorders that require medical detoxification will be initially excluded from participation, but will be eligible once they have completed their detoxification.
2. Veterans with comorbid Antisocial Personality Disorder, or history of animal cruelty will be excluded. Veterans with comorbid disorders that fall into the following DSM-5 categories will also be excluded: delirium, dementia, amnestic disorders, other cognitive disorders and psychotic disorders. Veterans with active Bipolar I or II and are not on a stable medication regime will be excluded.
3. Given evidence suggesting that benzodiazepine medications restrict the therapeutic benefits of PE, potential participants will be required to taper and cease use under supervision of their prescribing physician. Participants must be off benzodiazepines for at least two weeks prior to enrolling in the study. Patients using antidepressant medication for PTSD will be eligible for participation as long as they are on a stable regimen (i.e., consistent dose for at least two weeks prior to enrollment and throughout the study).
4. For safety purposes, Veterans who based on history or mental status examination have a significant risk of committing suicide, or who are homicidal or violent and who are in the Investigator's opinion in significant imminent risk of hurting others, will be excluded.
5. Patients who are unable to speak, read, and understand English or are judged by the investigator to be unable or unlikely to follow the study protocol and complete all scheduled visits.
6. Patients who report a dog phobia or are otherwise opposed to working with dogs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Emotional Numbing Symptoms of PTSD | Through therapy completion (an average of 12 weeks)
  Clinician Administered PTSD Scale (CAPS) clinical interview - Emotional Numbing Item
Change in Emotional Numbing Symptoms of PTSD | Through therapy completion (an average of 12 weeks)
  Posttraumatic Stress Disorder Checklist (PCL) self-report questionnaire -

SECONDARY OUTCOMES:
Change in Treatment Engagement | Through therapy completion (an average of 12 weeks)
  Number of therapy sessions attended
Change in PTSD diagnosis - interview | Through therapy completion (an average of 12 weeks)
  No longer meeting diagnostic criteria for PTSD via the Clinician Administered PTSD scale (CAPS) clinical interview
Change in PTSD diagnosis - self-report | Through therapy completion (an average of 12 weeks)
  No longer meeting diagnostic criteria for PTSD via self-report PTSD symptoms on the PTSD Checklist (PCL)

CONTACTS AND LOCATIONS:
Overall Officials: Anouk Grubaugh, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center
Locations (1):
- Ralph H. Johnson VAMC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grubaugh AL, Myers US, Keller SM, Wangelin BC, Lozano BE, Tuerk PW. An adjunctive human-animal interaction intervention for veterans with PTSD: study protocol for a randomized controlled trial. Trials. 2019 Dec 27;20(1):786. doi: 10.1186/s13063-019-3877-3. PMID 31881993